CLINICAL TRIAL: NCT02236884
Title: A Pilot Study of the Feasibility and Safety of No-scar Transanal Total Mesorectal Excision for Rectal Cancer Without Conventional Laparoscopic Assistance
Brief Title: The Feasibility and Safety of No-scar Transanal Total Mesorectal Excision for Rectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, doctor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIHSYSU08; D2014002 (Other: sysu 6th hospital)
Record Dates: First submitted 2014-09-04; First posted 2014-09-11 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2014-09

CONDITIONS: Rectal Cancer; Surgery
Keywords: rectal cancer; no scar; NOTES; TaTME; feasibility; safety
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- no-scar transanal TME (Experimental): no-scar transanal total mesorectal excision(TME) of rectal cancer
  Interventions: Procedure: no-scar transanal total mesorectal excision(TME)

INTERVENTIONS:
Procedure: no-scar transanal total mesorectal excision(TME)
  Other Names: Pure NOTES transanal TME; TaTME; TAMIS TME; single-port transanal TME

SUMMARY:
During the past three years, a revolutionized radical surgical approach for rectal cancer ("down to up TME " approach or "transanal TME (TaTME)"approach, which is opposite to the conventional approach) has emerged and it is a concept that combines natural orifice transluminal endoscopic surgery(NOTES) and total mesorectal excision(TME) with curative intent. The feasibility, safety and reproducibility of it were first demonstrated in swine survival experiments and subsequently in human cadaver series, and then it was successfully applied to human patients in few centers around the world, most of which were performed with assistance of laparoscopy, namely hybrid transanal TME. In addition, pure-NOTES without conventional laparoscopic assistance (no scar) has also been demonstrated, though the cases were more limited. In the initial stage, our group has successfully performed this no-scar transanal TME in a series of human cadavers with satisfactory outcome. Hence the investigators conduct this study, looking to see if this pure transanal NOTES investigational procedure is a safe and effective approach to radically remove rectal cancer of the mid and lower rectum and meanwhile, if it can reduce pain, gain faster recovery and better function and life quality when gaining the best cosmetic effect.

DETAILED DESCRIPTION:
Transanal total mesorectal excision (TaTME) is a novel development in the field of colorectal surgery which combines the mini-invasive concept of natural orifice transluminal endoscopic surgery(NOTES), the technique of single-port laparoscopic surgery and the principle of total mesorectal excision with curative intent for treating rectal cancer. Based on the platform of either transanal endoscopic microsurgery(TEM) or transanal minimally invasive surgery (TAMIS), it is an innovative way of retrograde TME dissection from bottom to up with or without laparoscopic assistance. It is supposed to facilitate distal rectal mobilization, thus achieving precise and sufficient distal margin and to reduced need for multiple stapler firings in transecting the rectum, consequently decreasing anastomotic leakage rates which is especially important for obese male patients with a narrow pelvis where exposure to the distal rectum from the abdominal approach can prove difficult. It could also protect neurovascular bundle with better visualization and exposure and has the advantage of better function and avoiding sacrificing sphincter. After a series of preclinical trail of animal and cadaver, it has been successfully applied to humans and successional reports have proved its feasibility and safety. However, the majority of published series is hybrid NOTES, which need the assistance of conventional laparoscopic surgery from above to bottom and abdominal incision, scar, pain and incision related complications such as wound infection, abscess, hernia and implanted incisional tumors cannot be necessary avoided. It is also worried that the cost will increased since two groups of surgical equipment are needed(the abdominal and perineal) and more surgical staff are required if the two team operate at the same time(two-team approach). Up to date, as far as we have known, the pure transanal TME NOTES without any laparoscopic assistance has also been successfully performed in human patients though the cases are rare. The investigators of our center have also successfully performed pure-NOTES rectal resection in human cadavers in the past few months, and are confident to move this forward to conduct this pilot study to evaluate the feasibility and safety of this surgery in rectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven adenocarcinoma of the rectum
* No previous abdominal surgery, no distant metastasis or synchronous colon cancer
* BMI≤ 35kg/m2
* Clinical staging (T1 or T2 or T3) with N1-2M0
* Patients of rectal adenocarcinoma with T3N0 or N (+) received preoperative concurrent chemoradiotherapy (CCRT) as neoadjuvant therapy
* Rectal cancer located 4-12 cm from the anal verge
* The diameter of primary tumor should <6cm
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* American Society of Anesthesiology (ASA) classⅠ to Ⅲ lesions
* After the evaluation of Multi-disciplinary team (MDT)
* Written informed consent

Exclusion Criteria:

* T4 tumor that invade the external sphincter or levator ani muscle or neighbor organs
* Recurrent rectal cancer
* Distant metastasis
* Obstructing rectal cancer
* Synchronous colon cancer
* Pregnant or breast-feeding women
* Fecal incontinence
* History of prior colorectal cancer
* History of inflammatory bowel disease
* Other malignancies diagnosed within the previous year
* Mental illness
* Any evidence of active infection
* History of bleeding diathesis or coagulopathy
* Impaired renal or hepatic function that could not tolerate surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Composite mesure of prioperative feasibility and safety | one-year
  To evaluate the feasibility and safety by operative time, estimated blood loss, intraoperative complications, convert to Hybrid NOTES or open surgery, pathological outcome including Total Mesorectal Excision (TME) quality, the lymph nodes harvested, and specimen length, circumferential margin, etc. and postoperative complications graded according to Clavien-Dindo, reoperation rate, 30-day mortality, 30-day readmission

SECONDARY OUTCOMES:
composite measure of life quality | 1-3 year
  To evaluate bladder function, anal function, sexual function and life quality by incontinence score, EORTC QLQ C30 and EORTC QLQ CR38, etc
Composite mesure of postoperative outcome | one-year
  To evaluate the postoperative outcome by length of hospital stay after operation, the time of first flatus, the time of recover to flow diet, postoperative pain by VAS, analgesic use ,etc
Composite mesure of oncological outcome | 1-3 year
  3-year disease free survival (DFS), 3-year local recurrence rate, 3-year distal metastasis rate, 3-year overall survival (cancer related or non-cancer related)

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Wang, MD, Study Director — Sun Yatsen University
Locations (1):
- Gastrointestinal Hospital, Sun Yatsen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Chen WH, Kang L, Luo SL, Zhang XW, Huang Y, Liu ZH, Wang JP. Transanal total mesorectal excision assisted by single-port laparoscopic surgery for low rectal cancer. Tech Coloproctol. 2015 Sep;19(9):527-34. doi: 10.1007/s10151-015-1342-1. Epub 2015 Jul 29. PMID 26220109
- [Result] Kang L, Chen WH, Luo SL, Luo YX, Liu ZH, Huang MJ, Wang JP. Transanal total mesorectal excision for rectal cancer: a preliminary report. Surg Endosc. 2016 Jun;30(6):2552-62. doi: 10.1007/s00464-015-4521-2. Epub 2015 Aug 27. PMID 26310534